CLINICAL TRIAL: NCT02600195
Title: Reduction of Infection in Neonatal Intensive Care Units Using the Evidence-based Practice for Improving Quality: A Cluster Randomised Trial
Brief Title: Reduction of Infection in Neonatal Intensive Care Units Using the Evidence-based Practice for Improving Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: China Medical Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-194
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Nosocomial Infections
Keywords: Intensive Care, Neonatal; Nosocomial Infections; Quality Improvement
MeSH Terms: conditions — Cross Infection | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPIQ sites (Experimental): Use Evidence-based Practice for Improving Quality (EPIQ) method to develop and implement evidence-based practice changes to reduce hospital-acquired infection
  Interventions: Behavioral: Evidence-based Practice for Improving Quality (EPIQ) method
- Control sites (No Intervention): Continue current practices

INTERVENTIONS:
Behavioral: Evidence-based Practice for Improving Quality (EPIQ) method — The intervention NICUs (n = 12) will receive training in the Evidence-based Practice for Improving Quality (EPIQ) method and then develop, implement, and document evidence-based practice changes to reduce hospital-acquired infection. Compliance with practice changes and neonatal outcomes will be monitored. NICUs will receive quarterly feedback on their progress, as well as access to implementation support.
  Arms: EPIQ sites

SUMMARY:
This 4-year cluster randomized controlled trial aims to determine whether implementation of Evidence-based Practice for Improving Quality (EPIQ) method can reduce hospital-acquired infection in Chinese Neonatal Intensive Care Units (NICUs).

DETAILED DESCRIPTION:
Following randomization into two groups, the intervention NICUs (n = 12) will receive training in the EPIQ method and then develop, implement, and document evidence-based practice changes to reduce hospital-acquired infection. Compliance with practice changes and neonatal outcomes will be monitored. NICUs will receive quarterly feedback on their progress, as well as access to implementation support. Control NICUs (n = 12) will collect neonatal data and continue to provide standard care. Study subjects will be all preterm infants born at <34 weeks' gestation and admitted to participating NICUs during the trial (estimated n = 5,200 per year). Data analysis will be conducted to compare neonatal outcomes and health-care resources used between the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at <34 weeks' gestation
* Admitted to the participating NICUs within 7 days after birth
* Admitted to the participating NICUs between May 1, 2015 and April 30, 2018

Exclusion Criteria:

* Infants with major congenital anomalies
* Infants who are moribund on admission (a decision is made to provide only palliative care)

Max Age: 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15600 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-04 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of hospital-acquired infection | Three years
  Combined cases of following types of hospital-acquired infection: ventilation associated pneumonia, central line-associated blood stream infection (CLABSI), blood stream infections excluding CLABSI, urinary tract infections, meningitis, clinical sepsis

SECONDARY OUTCOMES:
Incidence of ventilation associated pneumonia | Three years
Incidence of central line-associated blood stream infection | Three years
Incidence of blood stream infection excluding CLABSI | Three years
Incidence of meningitis | Three years
Incidence of clinical sepsis | Three years
Incidence of urinary tract infections | Three years
Incidence of stage ≥2 necrotizing enterocolitis | Three years
Days on ventilation support | Three years
Days on total parenteral nutrition | Three years
Days on antibiotics | Three years
Days on inotropes | Three years
All cause mortality | Three years
Infection-related mortality | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Yun Cao, MD, PHD, Principal Investigator — Children's Hospital of Fudan University; Vibhuti Shah, MD, Msc, Principal Investigator — University of Toronto; Shoo K Lee, MD, PHD, Principal Investigator — University of Toronto; Weiping Wang, MD, PHD, Principal Investigator — Fudan University
Locations (24):
- China (24):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Children's Hospital, Beijing, Beijing Municipality
  - Fujian Maternity and Child Health Care Hospital, Fuzhou, Fujian
  - Gansu Maternity and Child Health Care Hospital, Lanzhou, Gansu
  - Shenzhen Maternity and Child Health Care Hospital, Shenzhen, Guangdong
  - Guangxi Maternity and Child Health Care Hospital, Nanning, Guangxi
  - Guiyang Children's Hospital, Guiyang, Guizhou
  - Children's Hospital of Hebei Province, Shijiazhuang, Hebei
  - Zhengzhou Children's Hospital, Zhengzhou, Henan
  - Hubei Maternity and Child Health Care Hospital, Wuhan, Hubei
  - Tongji Hospital Affiliated to Tongji Medical College, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Children's Hospital, Nanjing, Jiangsu
  - Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - Wuxi Maternity and Child Health Care Hospital, Wuxi, Jiangsu
  - Jiangxi Children's Hospital, Nanchang, Jiangxi
  - Jinan Children's Hospital, Jinan, Shandong
  - Qingdao Maternity and Child Health Care Hospital, Qingdao, Shandong
  - Shanxi Maternity and Child Health Care Hospital, Taiyuan, Shanxi
  - Shanxi Maternity and Child Health Care Hospital, Xian, Shanxi
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Second Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang
  - Shanghai First Maternity and Child Health Care Hospital, Shanghai

REFERENCES:
- [Background] Lee SK, Aziz K, Singhal N, Cronin CM, James A, Lee DS, Matthew D, Ohlsson A, Sankaran K, Seshia M, Synnes A, Walker R, Whyte R, Langley J, MacNab YC, Stevens B, von Dadelszen P. Improving the quality of care for infants: a cluster randomized controlled trial. CMAJ. 2009 Oct 13;181(8):469-76. doi: 10.1503/cmaj.081727. Epub 2009 Aug 10. PMID 19667033
- [Background] Zhou Q, Lee SK, Jiang SY, Chen C, Kamaluddeen M, Hu XJ, Wang CQ, Cao Y. Efficacy of an infection control program in reducing ventilator-associated pneumonia in a Chinese neonatal intensive care unit. Am J Infect Control. 2013 Nov;41(11):1059-64. doi: 10.1016/j.ajic.2013.06.007. Epub 2013 Sep 14. PMID 24041863
- [Background] Polin RA, Denson S, Brady MT; Committee on Fetus and Newborn; Committee on Infectious Diseases. Strategies for prevention of health care-associated infections in the NICU. Pediatrics. 2012 Apr;129(4):e1085-93. doi: 10.1542/peds.2012-0145. Epub 2012 Mar 26. PMID 22451712
- [Background] Fanaroff AA, Hack M, Walsh MC. The NICHD neonatal research network: changes in practice and outcomes during the first 15 years. Semin Perinatol. 2003 Aug;27(4):281-7. doi: 10.1016/s0146-0005(03)00055-7. PMID 14510318
- [Background] Horbar JD, Soll RF, Edwards WH. The Vermont Oxford Network: a community of practice. Clin Perinatol. 2010 Mar;37(1):29-47. doi: 10.1016/j.clp.2010.01.003. PMID 20363446
- [Derived] Peng W, Han J, Li S, Zhang L, Yang C, Guo J, Cao Y. The Association of Human Milk Feeding With Short-Term Health Outcomes Among Chinese Very/Extremely Low Birth Weight Infants. J Hum Lact. 2022 Nov;38(4):670-677. doi: 10.1177/08903344221078237. Epub 2022 Mar 2. PMID 35236170
- [Derived] Luo N, Jiang S, McNamara PJ, Li X, Guo Y, Wang Y, Han J, Deng Y, Yang Y, Lee SK, Cao Y. Cardiovascular Pharmacological Support Among Preterm Infants in Chinese Referral Center Neonatal Intensive Care Units. Front Pediatr. 2021 Apr 22;9:638540. doi: 10.3389/fped.2021.638540. eCollection 2021. PMID 33968845
- [Derived] Peng W, Jiang S, Li S, Xia S, Chen S, Yang Y, Lee SK, Cao Y. Human Milk Feeding Status of Preterm Infants in Neonatal Intensive Care Units in China. J Hum Lact. 2020 May;36(2):283-290. doi: 10.1177/0890334419901265. Epub 2020 Feb 20. PMID 32078781